CLINICAL TRIAL: NCT05363839
Title: A Phase 1, Single-center, Placebo-controlled, Double-blind, Randomized Trial to Assess the Safety, Tolerability, and Pharmacokinetics of Single Ascending Oral Doses of ACH-000029 in Healthy Subjects
Brief Title: To Assess the Safety, Tolerability and Pharmacokinetics of ACH-000029 in Healthy Subjects
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Based on the unblinded clinical data, the trial was terminated.
Sponsor: Syneos Health (Other)
Collaborators: Otsuka Pharmaceutical Development & Commercialization, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: X07-201-00001
Record Dates: First submitted 2022-03-01; First posted 2022-05-06 (Actual); Last update posted 2023-04-27 (Actual); Status verified 2023-01

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — ACH-000029

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SAD Cohorts 1 to 3 - Participants Receiving ACH-000029 (Experimental): Each SAD cohort participant will be randomized to receive 10mg for cohort 1; up to 30mg and up to 60mg for cohorts 2 and 3 respectively dependent on dose review committee.
  Interventions: Drug: ACH-000029
- SAD Cohorts 1 to 3 - Participants Receiving Placebo (Placebo Comparator): Each SAD cohort participant will be randomized to receive placebo on a ratio of 3:1 (active: placebo).
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ACH-000029 — ACH-000029 will be administered orally via a capsule.
  Arms: SAD Cohorts 1 to 3 - Participants Receiving ACH-000029
Drug: Placebo — Placebo will be administered orally via a capsule.
  Other Names: Matching Placebo
  Arms: SAD Cohorts 1 to 3 - Participants Receiving Placebo

SUMMARY:
Randomized single ascending dose placebo controlled treatment of ACH-000029 administered orally via capsule in healthy volunteers.

DETAILED DESCRIPTION:
This study will be conducted in up to 3 dosing groups of 8 total subjects each.

The purpose of this trial is to determine the safety and tolerability of a single dose of ACH-000029 or placebo.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or non-childbearing potential female.
* Surgically sterile male and female.

Exclusion Criteria:

* Breastfeeding female subjects.
* Clinical abnormal past medical history.
* History of drug and/or alcohol abuse within 2 years prior to screening.
* History of or current hepatitis or acquired immunodeficiency syndrome or carriers of hepatitis B surface antigen and/or anti-hepatitis C virus antibodies, or human immunodeficiency virus (HIV) antibodies.
* History of any significant drug allergy or known or suspected hypersensitivity.
* A positive urine or breath alcohol test and/or urine drug screen for substances of abuse at screening or upon admission to the trial site (Day -1).
* Subjects having taken an investigational drug within 30 days prior to screening or a biological investigational product within 30 days or 5 half-lives (whichever is longer) preceding screening, except the last dose of severe acute respiratory syndrome coronavirus (SARS-CoV-2 [COVID-19]) vaccine, which must be administered at least 7 days prior to screening.
* Any history of significant bleeding or hemorrhagic tendencies.
* Any history of difficulty in donating blood.
* The donation of blood or plasma within 30 days prior to the first dose of IMP.
* Use of prescription, over-the-counter, or herbal medications or vitamin supplements within 14 days prior to the first dose of IMP and oral antibiotics within 30 days prior to the first dose of IMP.
* Use of tobacco products or daily exposure to second-hand smoke within 2 months prior to the screening visit.
* Presenting with, or having a history of, uncontrolled hypertension (SBP > 140 mmHg or DBP > 90 mmHg) or symptomatic hypotension, or orthostatic hypotension, which is defined as a decrease of ≥ 30 mmHg in SBP or a decrease of ≥ 20 mmHg in DBP after at least 3 minutes of standing compared with the previous supine BP, OR development of symptoms.
* Supine HR, after resting for at least 3 minutes, outside the range of 50 to 90 bpm.
* Abnormal ECG findings at screening or check-in.
* History of unexplained syncope, where orthostatic likely event.
* Personal or family history of sudden death or long QT syndrome.
* History of serious mental disorders that, in the opinion of the investigator, would exclude the subject from participating in this trial.
* No permanent place of residence.
* Subjects with active suicidal ideation prior to dosing.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2022-05-06 (Actual); Primary Completion 2022-11-02 (Actual); Study Completion 2022-11-02 (Actual)

PRIMARY OUTCOMES:
Number (%) of subjects experiencing orthostatic hypotension at any timepoint | Screening (Days -28 to Day -2) to end of treatment Day 7
  Orthostatic assessment will be with the criteria ≥ 20 mmHg decrease in SBP and a > 25 bpm increase in HR from supine to standing.
Maximum change in timepoint-matched systolic blood pressure and diastolic blood pressure. | Screening (Days -28 to Day -2) to end of treatment Day 7
Maximum change in timepoint-matched resting heart rate. | Screening (Days -28 to Day -2) to end of treatment Day 7
Assessment of abnormal clinical laboratory tests (Hemoglobin & mean corpuscular hemoglobin concentration) | Screening (Days -28 to Day -2) to end of treatment Day 7
Assessment of abnormal clinical laboratory tests (Hematocrit) | Screening (Days -28 to Day -2) to end of treatment Day 7
Assessment of abnormal clinical laboratory tests (Mean corpuscular volume) | Screening (Days -28 to Day -2) to end of treatment Day 7
Assessment of abnormal clinical laboratory tests (RBC count) | Screening (Days -28 to Day -2) to end of treatment Day 7
Assessment of abnormal clinical laboratory tests (WBC count (absolute and differential)) | Screening (Days -28 to Day -2) to end of treatment Day 7
Assessment of abnormal clinical laboratory tests (Platelets) | Screening (Days -28 to Day -2) to end of treatment Day 7
Assessment of abnormal clinical laboratory tests (Mean platelet volume) | Screening (Days -28 to Day -2) to end of treatment Day 7
Assessment of abnormal clinical laboratory tests (Anion gap, bicarbonate, calcium, chloride, cholesterol, glucose, magnesium, potassium, sodium, creatinine, uric acid, triglycerides, urea) | Screening (Days -28 to Day -2) to end of treatment Day 7
Assessment of abnormal clinical laboratory tests (Lactate Dehydrogenase (LDH), Alanine Transaminase (ALT), gamma-glutamyl transferase (GGT), Alkaline phosphatase (ALP) , aspartate aminotransferase (AST), phosphatase, creatinine phosphokinase) | Screening (Days -28 to Day -2) to end of treatment Day 7
Assessment of abnormal clinical laboratory tests (Albumin) | Screening (Days -28 to Day -2) to end of treatment Day 7
Assessment of abnormal clinical laboratory tests (Glomerular filtration rate) | Screening (Days -28 to Day -2) to end of treatment Day 7
Assessment of abnormal clinical laboratory tests (Globulin) | Screening (Days -28 to Day -2) to end of treatment Day 7
Assessment of abnormal clinical laboratory tests (Total bilirubin) | Screening (Days -28 to Day -2) to end of treatment Day 7
Assessment of abnormal clinical laboratory tests (Total protein) | Screening (Days -28 to Day -2) to end of treatment Day 7
Coagulation | Screening (Days -28 to Day -2) to end of treatment Day 7
  Blood sample assessments will include activated partial thromboplastin time, prothrombin time-international normalized ratio.
Assessment of abnormal Urinalysis (Bilirubin, blood, glucose, ketones, nitrites, protein) | Screening (Days -28 to Day -2) to end of treatment Day 7
Assessment of abnormal Urinalysis (Leukocyte esterase) | Screening (Days -28 to Day -2) to end of treatment Day 7
Assessment of abnormal Urinalysis (Microscopic analysis) | Screening (Days -28 to Day -2) to end of treatment Day 7
Assessment of abnormal Urinalysis (pH) | Screening (Days -28 to Day -2) to end of treatment Day 7
Assessment of abnormal Urinalysis (Specific gravity) | Screening (Days -28 to Day -2) to end of treatment Day 7
Assessment of abnormal Vital signs (temperature) | Screening (Days -28 to Day -2) to end of treatment Day 7
  Temperature will be assessed after subject has been in supine position for at least 3 minutes.
Assessment of abnormal Vital signs (respiratory rate) | Screening (Days -28 to Day -2) to end of treatment Day 7
  Respiratory rate will be assessed after subject has been in supine position for at least 3 minutes.
Assessment of abnormal Vital signs (blood pressure) | Screening (Days -28 to Day -2) to end of treatment Day 7
  Blood pressure will be assessed in supine and standing positions in each position for at least 3 minutes.
Assessment of abnormal Vital signs (heart rate) | Screening (Days -28 to Day -2) to end of treatment Day 7
  Heart rate will be assessed in supine and standing positions in each position for at least 3 minutes.
Assessment of Physical examinations (height) | Screening (Days -28 to Day -2) to end of treatment Day 7
Assessment of Physical examinations (weight) | Screening (Days -28 to Day -2) to end of treatment Day 7
Assessment of Physical examinations (BMI) | Screening (Days -28 to Day -2) to end of treatment Day 7
Assessment of Physical examinations | Screening (Days -28 to Day -2) to end of treatment Day 7
  Subjects will be visually assessed for any abnormalities with head, eyes, ears, nose and throat; thorax; abdomen; urogenital; skin and mucosae.
Assessment of Neurological examinations | Screening (Days -28 to Day -2) to end of treatment Day 7
  Subjects will be assessed for any abnormalities and evaluated for mental status, cranial nerves, motor system, reflexes, sensory system, coordination and station and gait.
12-lead ECG assessment of PR interval | Screening (Days -28 to Day -2), Day -1, Day 1, Day 2, Day 4 and end of treatment Day 7
  Change in electrocardiograms
12-lead ECG assessment of QRS duration | Screening (Days -28 to Day -2), Day -1, Day 1, Day 2, Day 4 and end of treatment Day 7
  Change in electrocardiograms
12-lead ECG assessment of QT interval | Screening (Days -28 to Day -2), Day -1, Day 1, Day 2, Day 4 and end of treatment Day 7
  Change in electrocardiograms
12-lead ECG assessment of QTc | Screening (Days -28 to Day -2), Day -1, Day 1, Day 2, Day 4 and end of treatment Day 7
  Change in electrocardiograms
C-SSRS | Screening (Days -28 to Day -2) to end of treatment Day 7
  Subjects will be interviewed to capture the occurrence, severity and frequency of suicide-related thoughts and behaviors.
Monitoring of adverse events | Screening (Days -28 to Day -2) to end of treatment Day 7
  Any untoward medical occurrence in a subject, whether considered related to the treatment or not.
Pharmacokinetic assessment 1 | Day 1 to end of treatment Day 7
  Peak Plasma Concentration (Cmax)
Pharmacokinetic assessment 2 | Day 1 to end of treatment Day 7
  Time of peak plasma concentration (Tmax)
Pharmacokinetic assessment 3 | Day 1 to end of treatment Day 7
  Area under the concentration-time curve calculated to the last observable concentration at time (AUCt)
Pharmacokinetic assessment 4 | Day 1 to end of treatment Day 7
  Area under the concentration-time curve from zero to infinity (AUC∞)
Pharmacokinetic assessment 5 | Day 1 to end of treatment Day 7
  Apparent clearance of the drug normalized to body weight (CL/F)
Pharmacokinetic assessment 6 | Day 1 to end of treatment Day 7
  Apparent clearance of the drug normalized to body weight (CL/F)
Pharmacokinetic assessment 7 | Day 1 to end of treatment Day 7
  Terminal-phase elimination half-life (t1/2,z)
Pharmacokinetic assessment 8 | Day 1 to end of treatment Day 7
  Cmax normalized to dose (Cmax/Dose)
Pharmacokinetic assessment 9 | Day 1 to end of treatment Day 7
  Cmax normalized to dose (Cmax/Dose)
Pharmacokinetic assessment 10 | Day 1 to end of treatment Day 7
  AUCt normalized to dose (AUCt/Dose)
Pharmacokinetic assessment 11 | Day 1 to end of treatment Day 7
  AUC∞ normalized to dose (AUC∞/Dose)

CONTACTS AND LOCATIONS:
Locations (1):
- Nucleus Network Pty Ltd, Melbourne, Victoria, Australia

IPD SHARING:
Plan to Share IPD: No